CLINICAL TRIAL: NCT01864876
Title: A Randomized, Single-Blinded Phase 1 Study to Evaluate the Safety and Immunogenicity of a Single Administration of 5 mcg GLA in Healthy Volunteers
Brief Title: The Effects of GLA (5 mcg) on Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: MCA-0784
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — GLA-AF adjuvant; glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLA-AF (Experimental): 5 mcg GLA-AF given as one subcutaneous injection.
  Interventions: Biological: GLA-AF
- GLA-SE (Experimental): 5 mcg GLA-SE given as one intramuscular injection.
  Interventions: Biological: GLA-SE
- EM060G (SE) (Experimental): EM060G (SE) given as one intramuscular injection.
  Interventions: Biological: EM060G (SE)

INTERVENTIONS:
Biological: GLA-AF — Glucopyranosyl Lipid A (GLA) in an aqueous formulation (AF).
  Arms: GLA-AF
Biological: GLA-SE — Glucopyranosyl Lipid A (GLA) in a stable oil-in-water emulsion (SE).
  Arms: GLA-SE
Biological: EM060G (SE) — The same stable oil-in-water emulsion (SE), but without GLA.
  Arms: EM060G (SE)

SUMMARY:
This protocol is for a phase 1, randomized, single-blinded study to evaluate the safety and tolerability of a single 5 mcg dose of GLA-SE administered intramuscularly and GLA-AF administered subcutaneously. The second focus will be to detail the global immune response by measuring systemic cytokines, chemokines, and global gene regulation. The third focus will be to investigate the effects of GLA on the peripheral blood immune cells including monocytes and dendritic cells. The results of this trial will generate supportive human data to use GLA as an adjuvant in a dendritic cell-targeted vaccine strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females, as assessed by a medical history, physical exam,and laboratory tests;
2. Age of at least 18 years of age on the day of screening and no greater than 50 years at time of administration;
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 4 weeks);
4. Willing to undergo HIV testing and counseling and receive HIV test results;
5. If a female of child bearing potential, must be willing to use two effective methods of contraception (combined oral contraceptive pill; injectable contraceptive; diaphragm; Intra Uterine Device (IUD); condoms; anatomical sterility in self or partner) until 6 weeks after study drug administration. If a sexually active male, must be willing to use two effective methods of contraception (such as condoms, anatomical sterility) from screening until 6 weeks after study drug administration (same as above) and will be advised not to get his partner(s) pregnant during this time.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, positive for hepatitis C antibodies, or active syphilis infection based on clinical evaluation;
2. Confirmed HIV-1 or HIV-2 infection;
3. Any clinically significant abnormality on medical history or physical examination including history of immunodeficiency or autoimmune disease;
4. Any use of systemic corticosteroids immunosuppressive anticancer medications;
5. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation;
6. Any laboratory value outside of reference range other than CRP, with the exception of any non-clinically significant Grade I elevations of liver function tests (AST, ALT, direct/total bilirubin), electrolytes (Na, K, Cl, CO2), CBC, urinalysis as determined by the Principal Investigator or his designee.
7. Within the 12 months prior to enrollment, the subject self reports excessive daily alcohol use, frequent binge drinking or chronic marijuana abuse (defined as greater than 2 times a week) or any other use of illicit drugs;
8. If female, pregnant, planning a pregnancy during the trial period, or lactating;
9. Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days prior to study drug;
10. Prior receipt of GLA in another research study;
11. Participation in another clinical study of an investigational product currently or within past 16 weeks, or expected participation during this study;
12. In the opinion of the investigator, unlikely to comply with protocol due to medical, social or psychiatric reasons;
13. Allergy to eggs
14. A glomerular filtration rate that is less than 60 mL/min/1.73 m2 as calculated by study team based on laboratory creatinine values.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  Local reactogenicity events and systemic reactogenicity events will be monitored for 28 days post injection.
  * Local reactogenicity events include tenderness, erythema, skin discoloration, edema, vesicle formation or ulceration, induration, pruritus, formation of a crust or scab, or other.
  * Systemic reactogenicity events include fever, chills, headache, nausea, vomiting, malaise, myalgia, arthralgia, and rash.
  Long term safety will be monitored by follow-up phone calls at 3 months, 6 months, and 1 year post injection.

SECONDARY OUTCOMES:
Immunogenicity | 28 days
  Describe the global immune response by measuring systemic cytokines, chemokines and global gene regulation. Investigate the effects of GLA on the peripheral blood immune cells including monocytes and dendritic cells.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Rockefeller University, New York, New York, United States